CLINICAL TRIAL: NCT03667742
Title: SwEaTB - Diagnosing of Acute Tuberculosis
Brief Title: Diagnosing of Acute Tuberculosis
Acronym: SwEaTB
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01455; me17Eckstein2
Record Dates: First submitted 2018-08-22; First posted 2018-09-12 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Tuberculosis
Keywords: sweat protein markers in tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples, sweat samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: analysis of sweat and serum samples for protein markers — collection of blood and sweat samples (with Macroduct Sweat Collecting System) in patients with suspected tuberculosis or proven acute tuberculosis or pulmonary diseases (pneumonia, bronchitis, COPD) and analyzing serum and sweat for protein markers (Early Secretory Antigenic Target (ESAT-6) and Culture Filtrate Protein 10 (CFP-10) and C-reactive protein (CRP) and Amyloid A2 and complement component 1q (C1q)) by mass spectrometry and enzyme-linked immunosorbent assay (ELISA)

SUMMARY:
Sweat proteins are analysed to investigate differences in protein markers in patients with acute tuberculosis and other pulmonary diseases (pneumonia, Bronchitis, chronic obstructive pulmonary disease (COPD)) and healthy individuals. Differences in sweat protein markers in patients with positive and negative tuberculosis Enzyme-linked-immuno-Spot (EliSpot) are investigated.

Differences in sweat protein markers in the course of treatment in patients receiving tuberculostatic therapy are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Ability to understand the purpose of the study, provide signed and dated informed consent by patient or his/her legal representative
* In-patients with acute tuberculosis, suspected tuberculosis or other pulmonary diseases (pneumonia, Bronchitis, COPD)

Inclusion Criteria Healthy Donors:

* negative for Quantiferon- TB Gold Plus Test or ELISpot

Exclusion Criteria:

* Initiation of tuberculostatic therapy before baseline
* Initiation of antibiotic therapy in patients with other pulmonary diseases > 6 hours before baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 12 In- patients at University Hospital Basel/ Switzerland with acute tuberculosis 16 In- patients at University Hospital Basel/ Switzerland with other pulmonary diseases (Pneumonia, Bronchitis, COPD) 5 Healthy Donors
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Change in protein markers (ESAT-6 and CFP-10 and CRP and Amyloid A2 and C1q) in patients with tuberculosis and other pulmonary diseases | Sweat samples taken at baseline and 2 weeks after baseline
  Distinction of patients with acute tuberculosis from patients with other pulmonary diseases by protein markers (Early Secretory Antigenic Target (ESAT-6) and Culture Filtrate Protein 10 (CFP-10) and C-reactive protein (CRP) and Amyloid A2 and complement component 1q (C1q)). Analysis done by mass spectrometry and enzyme linked immunosorbent assay (ELIZA).
Change in protein markers (ESAT-6 and CFP-10 and CRP and Amyloid A2 and C1q) in patients with tuberculosis and other pulmonary diseases | Blood samples taken at baseline and 2 weeks after baseline
  Distinction of patients with acute tuberculosis from patients with other pulmonary diseases by protein markers (Early Secretory Antigenic Target (ESAT-6) and Culture Filtrate Protein 10 (CFP-10) and C-reactive protein (CRP) and Amyloid A2 and complement component 1q (C1q)). Analysis done by mass spectrometry and enzyme linked immunosorbent assay (ELIZA).

SECONDARY OUTCOMES:
change of protein markers during tuberculostatic therapy | sweat and blood sweat and blood samples taken at baseline and 2 weeks after initiating tuberculostatic therapy in patients with active tuberculosis
  Analysis of protein markers (Early Secretory Antigenic Target (ESAT-6) and Culture Filtrate Protein 10 (CFP-10) and C-reactive protein (CRP) and Amyloid A2 and complement component 1q (C1q)) during tuberculostatic therapy. Analysis done by mass spectrometry and enzyme linked immunosorbent assay (ELIZA).
Differences in protein markers in patients with other pulmonary diseases | sweat and blood samples taken at baseline
  Analysis and comparison of protein markers (Early Secretory Antigenic Target (ESAT-6) and Culture Filtrate Protein 10 (CFP-10) and C-reactive protein (CRP) and Amyloid A2 and complement component 1q (C1q)) in patients with other pulmonary diseases (pneumonia, Bronchitis, COPD). Analysis done by mass spectrometry and enzyme linked immunosorbent assay (ELIZA).
Differences in protein markers in patients with positive and negative tuberculosis ELISpot | sweat and blood samples taken at baseline
  Analysis and comparison of protein markers (Early Secretory Antigenic Target (ESAT-6) and Culture Filtrate Protein 10 (CFP-10) and C-reactive protein (CRP) and Amyloid A2 and complement component 1q (C1q)) in patients with positive and negative tuberculosis ELISpot. Analysis done by mass spectrometry and enzyme linked immunosorbent assay (ELIZA).

OTHER OUTCOMES:
detection of tuberculostatic drug in sweat samples in patients with active tuberculosis during tuberculostatic therapy | sweat samples taken 2 weeks after initiating tuberculostatic therapy in patients with active tuberculosis
  Analysis of sweat protein markers in patients with active tuberculosis during tuberculostatic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, PD Dr. med, Principal Investigator — Chief Clinical Medical Office
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Hochschule für Lifescience, Muttenz